CLINICAL TRIAL: NCT05893199
Title: Telemedicine in Atrial Fibrillation: Randomized Clinical Trial in Primary Care
Brief Title: Telemedicine in Atrial Fibrillation: Randomized Clinical Trial in Primary Care (AtrialConnect)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Domingo Orozco Beltrán, Professor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AtrialConnect
Record Dates: First submitted 2023-05-08; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
Keywords: Telemedicine; Atrial Fibrillation; Primary care; Patient perception; Quality of life; Efficacy; Efficiency; Job Satisfaction; Patient safety; Mobile Applications
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Patients in the intervention group (Telemedicine) will be followed up using the Ti.Care App in addition to the usual primary care follow-up.
  Interventions: Device: Clinical monitoring using the Ti.Care app (https://ti.care/es); Other: Usual care
- Primary care (Active Comparator): Patients in the control group will be followed up exclusively in primary care.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Clinical monitoring using the Ti.Care app (https://ti.care/es) — Clinical monitoring using the Ti.Care app (https://ti.care/es)
  Arms: Telemedicine
Other: Usual care — usual follow-up in primary care both arms

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia in the world, with a large consumption of health resources. Telemedicine represents a new model of care, facilitating the individual approach to each patient and reducing costs and complications.

This is an an open-label, randomized, multicenter, clinical trial aiming to analyze the use of telemedicine with AF patients in real clinical practice at primary care in terms of efficacy, efficiency, patient perception and professional satisfaction.

The intervention will be based on the use of the Ti.Care app as the telemedicine support, in addition to the usual care. The follow-up will be carried out for 12 months.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is the most common cardiac arrhythmia in the world, with a prevalence between 2-4%. Given the increase in prevalence, its associated morbidity and mortality, and the large consumption of health resources there has been a need to adapt health care models. Telemedicine and the use of mobile devices represent a new model of care for chronic patients, facilitating the individual approach to each patient and reducing the disability associated with their chronic pathology.

Objective: To analyze the use of telemedicine in patients with atrial fibrillation in real clinical practice in primary care trying in terms of efficacy (blood pressure control, incidence of ischemic stroke, incidence of bleeding), efficiency (number of visits to the clinic, hospitalizations, costs of care), patient perception (quality of life, therapeutic adherence, satisfaction with the mobile App) and professional satisfaction (satisfaction with the mobile App and benefits of its use in the clinic).

Methods: The investigators propose to conduct an open-label, randomized, multicenter clinical trial. The intervention will be based on the use of the Ti.Care app as the telemedicine support, in addition to the usual care with their primary care physician (PCP). The control group will perform the usual follow-up with their PCP. The follow-up will be carried out for 12 months, and is proposed as an effective and cost-efficient improvement for the national health system and for the patient.

Key words: Telemedicine, Mobile Applications, Atrial Fibrillation, Primary Health Care.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age diagnosed with AF.
* Without difficulties in using the mobile App or patients with difficulties in using the mobile App but with good family or caregiver support, who understand its use.

Exclusion Criteria:

* Terminally ill patient.
* Refusal to participate on the part of the patient
* Difficulties in understanding the contents of the mobile App (cognitive impairment, dependence for activities of daily living, etc.) and no enabling family support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | one year
  Measured with systolic and diastolic blood pressure
Incidence of ischemic stroke | one year
  Measured as the number of recorded ischaemic stroke events in the study months.
Incidence of bleeding | one year
  Number of bleeding events of any type recorded during follow-up.
Number of emergency visits | one year
  Number of recorded visits to the emergency department in the study months.
Number of hospitalizations | one year
  Number of hospital admissions for AF decompensation and its associated diseases during the study period.
Number of visits to primary care | one year
  Number of registered visits to the primary care service in the study months.
Costs of care | one year
  The indexes and prices of the Consejería de Sanidad for each type of consultation or hospitalisation and the established retail prices in the year of the study for medicines will be used.
Health-Related Quality Of Life | one year
  Measured with EuroQol 5D questionnaire
Therapeutic adherence | one year
  Measured with MMAS-8 Test (High adherence (8 or > 8 points), medium (6 or 7 points) and low adherence (5 or <5 points))
Patient satisfaction with the mobile application | one year
  Measured by the survey on satisfaction and perception of the use of new technologies in the field (designed for the study). Scoring: High satisfaction (4 or 5 points), medium (3 points), low satisfaction (1 or 2 points).
Professionals' satisfaction with the mobile application | one year
  Measured by the survey on satisfaction and perception of the use of new technologies in the field (designed for the study). Scoring: High satisfaction (5-7 points), medium (3 or 4 points), low satisfaction (1 or 2 points).

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Jordá Baldó, Medicine, Principal Investigator — Physician at Virgen del Puerto Hospital; Domingo L Orozco Beltrán, Medicine, Study Director — Professor at Miguel Hernández University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Result] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Result] Orozco-Beltran D, Brotons Cuixart C, Aleman Sanchez JJ, Banegas Banegas JR, Cebrian-Cuenca AM, Gil Guillen VF, Martin Rioboo E, Navarro Perez J. [Cardiovascular preventive recommendations. PAPPS 2020 update]. Aten Primaria. 2020 Nov;52 Suppl 2(Suppl 2):5-31. doi: 10.1016/j.aprim.2020.08.002. Spanish. PMID 33388118
- [Result] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Result] MacKinnon GE, Brittain EL. Mobile Health Technologies in Cardiopulmonary Disease. Chest. 2020 Mar;157(3):654-664. doi: 10.1016/j.chest.2019.10.015. Epub 2019 Oct 31. PMID 31678305
- [Result] Orozco-Beltran D, Sanchez-Molla M, Sanchez JJ, Mira JJ; ValCronic Research Group. Telemedicine in Primary Care for Patients With Chronic Conditions: The ValCronic Quasi-Experimental Study. J Med Internet Res. 2017 Dec 15;19(12):e400. doi: 10.2196/jmir.7677. PMID 29246881
- [Result] Pezel T, Berthelot E, Gauthier J, Chong-Nguyen C, Iliou MC, Juilliere Y, Galinier MC, De Groote P, Beauvais F, Bauer F, Vergeylen U, Gellen B, Raphael P, Bezard M, Ricci JE, Boiteux MC, Bonnefous L, Bodez D, Audureau E, Damy T. Epidemiological characteristics and therapeutic management of patients with chronic heart failure who use smartphones: Potential impact of a dedicated smartphone application (report from the OFICSel study). Arch Cardiovasc Dis. 2021 Jan;114(1):51-58. doi: 10.1016/j.acvd.2020.05.006. Epub 2020 Aug 28. PMID 32868257
- [Result] Herdman M, Badia X, Berra S. [EuroQol-5D: a simple alternative for measuring health-related quality of life in primary care]. Aten Primaria. 2001 Oct 15;28(6):425-30. doi: 10.1016/s0212-6567(01)70406-4. No abstract available. Spanish. PMID 11602124
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505